CLINICAL TRIAL: NCT01664039
Title: Assessing the Efficacy and Tolerability of TRAVATAN® Solution Without BAK, Containing Polyquad® Preservative (Travoprost 0.004%) Versus LUMIGAN® 0.01% Solution With BAK (Bimatoprost 0.01%) in Treatment Naïve Patients With Ocular Hypertension or Open Angle Glaucoma
Brief Title: An Efficacy and Tolerability Study of TRAVATAN® Versus LUMIGAN®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDG-11-244; 2012-002078-30 (EudraCT Number)
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2015-07-14 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Travoprost; Ophthalmic Solutions; Bimatoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRAVATAN (Experimental): Travoprost 0.004% ophthalmic solution with Polyquad®, 1 drop to the study eye(s), once a day in the evening, for 6 months
  Interventions: Drug: Travoprost 0.004% ophthalmic solution
- LUMIGAN (Active Comparator): Bimatoprost 0.01% ophthalmic solution with BAK, 1 drop to the study eye(s), once a day in the evening, for 6 months
  Interventions: Drug: Bimatoprost 0.01% ophthalmic solution

INTERVENTIONS:
Drug: Travoprost 0.004% ophthalmic solution — Ophthalmic solution without benzalkonium chloride (BAK), containing Polyquad® preservative
  Other Names: TRAVATAN®
  Arms: TRAVATAN
Drug: Bimatoprost 0.01% ophthalmic solution — Ophthalmic solution containing benzalkonium chloride (BAK)
  Other Names: LUMIGAN®
  Arms: LUMIGAN

SUMMARY:
The purpose of this study is evaluate effects of TRAVATAN® versus LUMIGAN® on intraocular pressure (IOP) and ocular surface and inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with either open-angle glaucoma or ocular hypertension in at least one eye and be treatment naïve to any glaucoma treatment.
* Intraocular pressure (IOP) between 19 mmHg and 35 mmHg in at least one eye, which would be the study eye.
* IOP considered to be safe (in the opinion of the investigator), in both eyes, in such a way that should assure clinical stability of vision and the optic nerve throughout the study period.
* Able to follow instructions and be willing and able to attend all study visits.
* Best corrected Snellen visual acuity of 6/60 (20/200, 1.0 LogMAR) or better in each eye.
* Must read, sign, and date an Ethics Committee-approved informed consent form.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known medical history of allergy, hypersensitivity or poor tolerance to any components of the study medications to be used in this study that is deemed clinically significant in the opinion of the Principal Investigator.
* Any abnormality preventing reliable applanation tonometry in either eye.
* Concurrent infectious/noninfectious conjunctivitis, keratitis or uveitis in either eye.
* Prior treatment of dry eye with punctal plugs, punctal cautery, Restasis® or topical ocular corticosteroids.
* History of ocular surface disease (dry eye) or current/prior use of dry eye medications (either over-the counter or prescription medications).
* Contact lens wear.
* Intraocular conventional surgery or laser surgery in either eye that is less than three months prior to the Screening Visit.
* Use of any systemic medications known to affect IOP (e.g., oral beta-adrenergic blockers, alpha-agonists and blockers, angiotensin converting enzyme inhibitors and calcium channel blockers), which have not been on a stable course for at least 7 days prior to Screening Visit or an anticipated change in the dosage during the course of the study.
* Women of childbearing potential not using reliable means of birth control, are pregnant, or lactating.
* Unwilling to risk the possibility of darkened iris or eyelash changes.
* Participation in any other investigational study within 30 days prior to the Screening Visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 2 study centers located in Slovenia.
Pre-assignment Details: All enrolled subjects were randomized. This reporting group includes all randomized subjects (104). Note: 1 subject randomized to Travatan and 3 subjects randomized to Lumigan did not receive treatment.
Groups:
- TRAVATAN: One drop to the study eye(s) once a day in the evening for 6 months
- LUMIGAN: One drop to the study eye(s) once a day in the evening, for 6 months
Period: Overall Study
Arm/Group | TRAVATAN | LUMIGAN
Started | 52 | 52
Completed | 46 | 43
Not Completed | 6 | 9
Not completed — Adverse Event | 3 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Noncompliance | 1 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects.
Groups:
- LUMIGAN: One drop to the study eye(s) once a day in the evening for 6 months
- Total: Total of all reporting groups
Arm/Group | TRAVATAN | LUMIGAN | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Customized [Number; unit: participants]
  Under 60 years | 25 | 26 | 51
  60 or more years | 27 | 26 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 16 | 51
  Male | 17 | 36 | 53

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Intraocular Pressure (IOP) at Month 6
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and measured in millimeters of mercury (mmHg). A more negative change indicates a greater amount of improvement. One eye was chosen as the study eye, and only data from the study eye were used for the analysis.
Time Frame: Baseline (Day 0), Month 6
Population: This analysis population includes all randomized subjects who received at least 1 dose of either study treatment and had at least 1 post-baseline on therapy study visit. Here, "n" is the number of subjects with non-missing values at the specific time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | TRAVATAN | LUMIGAN
Number analyzed (Participants) | 50 | 49
mmHg
  Baseline (Day 0) | 24.66 (3.65) | 24.59 (4.14)
  Change from Baseline at Month 6, n=46,43 | -7.61 (4.32) | -7.35 (3.84)

2. Secondary Outcome: Mean Change From Baseline in IOP at Week 6 and Month 3
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and measured in mmHg. A more negative change indicates a greater amount of improvement. One eye was chosen as the study eye, and only data from the study eye were used for the analysis.
Time Frame: Baseline (Day 0), Week 6, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | TRAVATAN | LUMIGAN
Number analyzed (Participants) | 50 | 49
mmHg
  Change from Baseline at Week 6, n=46,46 | -7.50 (3.80) | -7.02 (3.28)
  Change from Baseline at Month 3, n=46,44 | -7.96 (3.71) | -7.82 (3.15)

3. Secondary Outcome: Percentage of Subjects Who Reached Target IOP at Each Visit
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and measured in mmHg. Target IOP was defined as ≤ 18 mmHg. One eye was chosen as the study eye, and only data from the study eye were used for the analysis.
Time Frame: Week 6, Month 3, Month 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | TRAVATAN | LUMIGAN
Number analyzed (Participants) | 50 | 49
percentage of participants
  Week 6, n=46,46 | 69.6 | 56.5
  Month 3, n=46,44 | 71.7 | 70.5
  Month 6, n=46,43 | 73.9 | 67.4

4. Secondary Outcome: Number of Subjects With Change From Baseline in Ocular Hyperaemia by Grade at Each Visit
Description: Ocular Hyperaemia (excess of blood in the white of the eyes (sclera)) was graded by the investigator on a 4-point scale where 0=None/Trace, 1=Mild, 2=Moderate, and 3=Severe. One eye was chosen as the study eye, and only data from the study eye were used for the analysis.
Time Frame: Baseline (Day 0), Week 6, Month 3, Month 6
Population: This analysis population includes all randomized subjects who received at least 1 dose of either study treatment and had at least 1 post-baseline on therapy study visit with non-missing values by grade at the specific time point.
Measure: Number; unit: participants
Arm/Group | TRAVATAN | LUMIGAN
Number analyzed (Participants) | 50 | 49
participants
  Baseline, Grade 0 | 40 | 31
  Baseline, Grade 1 | 9 | 17
  Baseline, Grade 2 | 1 | 1
  -1 Grade Change from Baseline at Week 6 | 2 | 1
  0 Grade Change from Baseline at Week 6 | 20 | 23
  +1 Grade Change from Baseline at Week 6 | 23 | 20
  +2 Grade Change from Baseline at Week 6 | 1 | 2
  -1 Grade Change from Baseline at Month 3 | 2 | 1
  0 Grade Change from Baseline at Month 3 | 13 | 15
  +1 Grade Change from Baseline at Month 3 | 25 | 26
  +2 Grade Change from Baseline at Month 3 | 6 | 2
  -1 Grade Change from Baseline at Month 6 | 0 | 1
  0 Grade Change from Baseline at Month 6 | 20 | 15
  +1 Grade Change from Baseline at Month 6 | 23 | 25
  +2 Grade Change from Baseline at Month 6 | 3 | 2

5. Secondary Outcome: Number of Subjects With Change From Baseline in Corneal Staining by Grade at Month 3 and Month 6
Description: Corneal staining was assessed after ophthalmic dye was instilled in the eye. The upper eyelid was lifted slightly, and the eye was compared to grading panels. Corneal staining was graded on a scale from 0 (absent) to 5 (severe). One eye was chosen as the study eye, and only data from the study eye were used for the analysis.
Time Frame: Baseline (Day 0), Month 3, Month 6
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | TRAVATAN | LUMIGAN
Number analyzed (Participants) | 50 | 49
participants
  Baseline, Grade 0 | 41 | 39
  Baseline, Grade 1 | 8 | 9
  Baseline, Grade 2 | 1 | 1
  -1 Grade Change from Baseline at Month 3 | 7 | 4
  0 Grade Change from Baseline at Month 3 | 33 | 33
  +1 Grade Change from Baseline at Month 3 | 6 | 7
  -1 Grade Change from Baseline at Month 6 | 4 | 7
  0 Grade Change from Baseline at Month 6 | 28 | 25
  +1 Grade Change from Baseline at Month 6 | 13 | 10
  +2 Grade Change from Baseline at Month 6 | 1 | 1

6. Secondary Outcome: Number of Subjects With Change From Baseline in Conjunctiva Staining by Grade at Month 3 and Month 6
Description: Conjunctiva staining was assessed after ophthalmic dye was instilled in the eye. The upper eyelid was lifted slightly, and the eye was compared to grading panels. Conjunctiva staining was graded on a scale from 0 (absent) to 5 (severe). One eye was chosen as the study eye, and only data from the study eye were used for the analysis.
Time Frame: Baseline (Day 0), Month 3, Month 6
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | TRAVATAN | LUMIGAN
Number analyzed (Participants) | 50 | 49
participants
  Baseline, Grade 0 | 44 | 39
  Baseline, Grade 1 | 6 | 9
  Baseline, Grade 2 | 0 | 1
  Month 3, -1 Grade Change from Baseline | 6 | 6
  Month 3, 0 Grade Change from Baseline | 36 | 33
  Month 3, +1 Grade Change from Baseline | 3 | 5
  Month 3, +2 Grade Change from Baseline | 1 | 0
  Month 6, -1 Grade Change from Baseline | 4 | 7
  Month 6, 0 Grade Change from Baseline | 31 | 26
  Month 6, +1 Grade Change from Baseline | 11 | 9
  Month 6, +2 Grade Change from Baseline | 0 | 1

7. Secondary Outcome: Mean Change From Baseline in Ocular Surface Disease Index (OSDI) Score at Month 3 and Month 6
Description: The OSDI questionnaire (used to measure vision-related function, ocular symptoms, visual function, and environmental factors that may affect vision) was answered by the subject. Each of the 12 items was scored on a 0-4 Likert scale, where 0 is "None of the time" and 4 is "All of the time." A resultant overall 0-100 score was calculated, with higher scores representing greater disability. A negative number change represents a perceived improvement in ocular health.
Time Frame: Baseline (Day 0), Month 3, Month 6
Population: This analysis population includes all randomized subjects who completed the questionnaire at baseline, received at least 1 dose of either study treatment, and had at least 1 post-baseline on-therapy study visit. Here, "n" is the number of subjects with non-missing values at the specific time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TRAVATAN | LUMIGAN
Number analyzed (Participants) | 48 | 48
units on a scale
  Baseline (Day 0) | 14.6 (14.8) | 10.6 (10.5)
  Change from Baseline at Month 3, n=44,43 | -0.3 (12.2) | 0.0 (10.4)
  Change from Baseline at Month 6, n=44,42 | 0.4 (16.2) | 1.7 (14.3)

8. Secondary Outcome: Mean Change From Baseline In Tear Film Break Up Time (TBUT) at Month 3 and Month 6
Description: TBUT (the time required for dry spots to appear on the corneal surface after blinking) was assessed by the investigator using slit lamp examination . A longer break up time is a sign of a more stable tear film. A positive number change from baseline indicates improvement. One eye was chosen as the study eye, and only data from the study eye were used for the analysis.
Time Frame: Baseline (Day 0), Month 3, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | TRAVATAN | LUMIGAN
Number analyzed (Participants) | 50 | 49
seconds
  Baseline (Day 0) | 10.7 (2.7) | 11.7 (3.2)
  Change from Baseline at Month 3, n=46,44 | -1.6 (5.3) | -1.8 (4.0)
  Change from Baseline at Month 6, n=46,43 | -2.2 (3.6) | -2.2 (5.1)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (Sep 2012 - Jun 2014). This analysis population includes all subjects who received at least 1 dose of either study treatment.
Description: An AE was defined as any untoward medical occurrence in a patient who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. AEs were obtained as both volunteered and elicited comments from the study subjects.
Arm/Group | TRAVATAN | LUMIGAN
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/49
Other Adverse Events (participants affected / at risk) | 0/51 | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TRAVATAN (N=51) | LUMIGAN (N=49)
Thromboendarterectomy (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.